CLINICAL TRIAL: NCT05444400
Title: Acute Effects of Strengthening the Lower Limbs on Physical Function and Pain in Patients Operated on by Total Knee Arthroplasty
Brief Title: Acute Effects of Strengthening Lower Limbs Operated by Total Knee Arthroplasty
Acronym: AESLLKNEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Laura López-Bueno, Director Laura López-Bueno, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID0003
Record Dates: First submitted 2022-06-21; First posted 2022-07-05 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strengthening of lower limbs (Experimental): The participants of this group will carry out their training following the protocol described. The participants work with strength of lower limbs.
  Interventions: Other: Strengthening
- Conventional protocol (Active Comparator): The participants of this group will carry out their rehabilitation following the conventional protocol.
  Interventions: Other: Conventional protocol

INTERVENTIONS:
Other: Strengthening — Strengthening
  Arms: Strengthening of lower limbs
Other: Conventional protocol — Conventional protocol
  Arms: Conventional protocol

SUMMARY:
Knee osteoarthritis is a chronic joint disease and one of the leading causes of disability among adults, resulting in irreversible damage to articular cartilage and subchondral bone, osteophyte formation, joint pain and stiffness.The purpose of the study is to evaluate the acute responses of lower limb strengthening on physical function and pain, in patients operated on by total knee arthroplasty.Candidates for this study will be men and women over 55 years of age who have undergone total knee arthroplasty, who are admitted to the University Clinical Hospital of Valencia, with an intervention date in 2022-2023, and who begin their physiotherapy treatment between days 1-2 post-surgical.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a chronic joint disease and one of the leading causes of disability among adults, resulting in irreversible damage to articular cartilage and subchondral bone, osteophyte formation, joint pain and stiffness. Knee osteoarthritis often makes it difficult to participate in activities of daily living, which can make work difficult or even impossible, especially when it comes to physical activities that impose a great mechanical strain on the knee. For example, when climbing stairs, the pressure on the knees is six times greater than body weight, which is a known risk factor for knee OA due to occupational activities.Given the increasing prevalence of knee OA with the ageing population and the increasing state retirement age in most European countries, the implications of knee OA need to receive special attention.The most common surgical solution is the placement of a total knee arthroplasty, There are several reasons why your doctor might recommend knee replacement surgery. Recommendations for surgery are based on the patient's pain and disability, not age. Most patients who undergo a total knee replacement are between the ages of 55 and 80, but orthopedic surgeons evaluate patients individually. Usually, the surgical procedure takes between 1 and 2 hours. The orthopedic surgeon will remove the damaged cartilage and bone, and then place the new metal and/or plastic implants to restore knee alignment and function.The purpose of the study is to evaluate the acute responses of lower limb strengthening on physical function and pain, in patients operated on by total knee arthroplasty. Candidates for this study will be men and women over 55 years of age who have undergone total knee arthroplasty, who are admitted to the University Clinical Hospital of Valencia, with an intervention date in 2022-2023, and who begin their physiotherapy treatment between days 1-2 post-surgical. Patients will voluntarily participate in the study. All of them will be informed about the objectives and content of the research and written informed consent will be obtained. The study will conform to the Declaration of Helsinki and will be approved by the local ethics committee.Participants will be excluded if they have any involvement in the contralateral lower limb, if they have already had/have any other knee injury or other anatomical part of the intervened MI (in the last year), and if they have any other condition or disease in which there is a contraindication to physical exercise. Also if they participate in other research studies. In addition, if severe neural or vascular injury is evident.In a previous study, initial WOMAC scores had a standard deviation of 11. If the difference between the means of the intervention and control groups is at least 10, a sample size of 20 patients in each group is adequate to reject the null hypothesis with a power of 80% and a significance level of p < 0.05.If possible, two days before the surgical intervention, a video will be sent to the participants with the performance of the exercises to be performed, so that they can check the technique to be executed. Likewise, they will be sent the following information about guidelines to follow for the realization of the tests:

• Try to rest at least 8 hours the post-surgical night. Patients will be treated while admitted to the hospital (between 3 and 4 days), through 1 session / day of approximately 40 minutes.

Evaluation 1 will be performed on the first day after surgery (1st postoperative day) and evaluation 2 on the day of hospital discharge (3rd postoperative day).EXERCISE PROGRAM WITH ELASTIC RESISTANCE:

* All exercises are done until the maximum number of repetitions is reached, since they will only be done once / day.
* During the first day, each exercise should begin with 2 sets of 2 repetitions as a warm-up and calculation of the appropriate intensity. The appropriate intensity will be the one where the patient tells us that he perceives 5-6 out of 10 on the Borg CR10 scale after finishing 2 repetitions.CONTROL GROUP EXERCISE PROGRAM:

The patients of the control group will perform the physiotherapy exercises following the RHB protocol in ATR of the University Clinical Hospital of Valencia.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 55 years of age.
* Total knee arthroplasty
* Intervention date in 2022, and who begin their physiotherapy treatment between days 1-2 post-surgical.

Exclusion Criteria:

* Participants have any involvement in the contralateral lower limb.
* Participants have already had/have any other knee injury or other anatomical part of the intervened LM (in the last year).
* Participants have any other condition or disease in which there is a contraindication to physical exercise.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Strength | 3 days
  Number of repetitions achieved in each day and exercise. REGISTRO DE....

SECONDARY OUTCOMES:
Kinesiophobia | 3 days
  Kinesiophobia will be evaluated (REPASAR) mainly through the Spanish version of the Kinesiophobia Tampa Scale in a selfrecorded manner.
Pain intensity | 3 days
  The patient will be mark a point on the scale and subsequently, the clinician or researcher quantifies the number of mm indicated by the patient. The level is from 0 to 100 mm.
Pain percepcion | 3 days
  The chronic pain perception will be measured by Questionnaire on Perception of Self-Efficacy in the Face of Chronic Pain (CPSS) that contains 19 items and evaluates 3 domains: self-efficacy for pain management (α=0.72), physical functioning (α=0.98) and symptom management (α=0.85).
Range of motion | 3 days
  The degrees of movement (ROM) of the following joints shall be actively and passively measured by means of a manual goniometer.
Isometric knee extension/flexion force | 3 days
  They will be evaluated with a portable handheld dynamometer.maximum contractions of 5 seconds will be performed, separated by 1 minute of rest, selecting the average value of these 3 for later analysis.
Self-administered physical function | 3 days
  WOMAC questionnaire be used to assess stiffness, pain and physical function in a self-administered manner. The questionnaire is a multidimensional scale composed of 24 items divided into 3 domains: functional pain (5 items), stiffness (2 items) and difficulties in activities of daily living (17 items).
Catastrophism | 3 days
  Scale of Catastrophism before pain in a self-registered way, which consists of 13 items that describe different thoughts and feelings associated with pain. The scale has 5 degrees, being 0 nothing at all, 1 a little, 2 moderately, 3 a lot and 4 all the time. The subject must mark his situation in each case. The scale consists of 13 items in total (0-52 points). Higher scores will indicate higher levels of pain catastrophism.
Perceived change | 3 days
  From the beginning of the study (first day after the operation), my general physical condition will be measure by Patients Global Impression Change (PGIC). The level is from 1 (I have improved a lot) to 7 (I have gotten a lot worse).
Gait functionality | 3 days
  The Time up and go (TUG) measures the time it takes for a person to get up from a standard chair (without using their arms to get up), walk to a line on the floor 3m away, turn around, walk back to the chair, and sit down again. Walking aids (e.g. walker) are allowed if necessary. Two tests are performed, with one minute of rest between them, using the highest value for analysis.
Spillage from the knee joint | 3 days
  It was assessed by measuring knee circumference. Patients lie on a stretcher with the operated knee relaxed and extended as much as possible. If the knee can extend below 0°, a cylinder is placed under the heel. A non-elastic tape measure was carefully placed and adjusted 1 cm above the base of the kneecap. Knee joint circumference was measured twice and the highest value was used for analysis.
Pressure pain thresholds | 3 days
  UDP is defined as the minimum amount of pressure in which a feeling of pressure is transformed into a sensation of pain. The mechanical pressure instrument, called an algometer (Wagner Instruments, Greenwich, CT, USA), will be used in this study. This consists of a round rubber disc (1 cm2 in surface) attached to a pressure (force)
Use of analgesics | 3 days
  we assessed the number of days on which participants were taking painkillers during the week. The following question was asked of the participants: "As a result of the pain, how many days during this week did you take painkillers?" Participants had to respond with a number of 0-7, and the drugs administered were recorded in the hospitalization room.

CONTACTS AND LOCATIONS:
Locations (1):
- Laura López-Bueno, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nunez-Cortes R, Lopez-Bueno L, Lopez-Bueno R, Cuenca-Martinez F, Suso-Marti L, Silvestre A, Casana J, Cruz-Montecinos C, Andersen LL, Calatayud J. Acute Effects of In-Hospital Resistance Training on Clinical Outcomes in Patients Undergoing Total Knee Arthroplasty: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2024 May 1;103(5):401-409. doi: 10.1097/PHM.0000000000002366. Epub 2023 Nov 22. PMID 38063321